CLINICAL TRIAL: NCT03486626
Title: Endometrial Thickness And Subendometrial Vascularity In Anovulatory Polycystic Ovarian Syndrome Patients Treated by Metformin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Adel mohamed kamal Eldin Abdelrahman, Resident of Obstetrics and gynecology, Ain Shams Maternity Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ain ShamsMH
Record Dates: First submitted 2018-03-25; First posted 2018-04-03 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Polycystic Ovary Syndrome; Anovulatory
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin to increase pregnancy rate in polycystic ovarian syndrome patients

SUMMARY:
The participants will receive metformin 500mg 3times per day for 3months and one month is left for spontaneous pregnancy to occur or not (primary outcome ) and the investigators will check endometrial thickness and subendometerial vascularity as markers of endometrial receptivity before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* PCO syndrome patients have the following criteria:

Age of the patient between 20 - 40 years old. All subjects are not on a specific diet nor a certain program of physical exercise Complaining of infertility either primary or secondary due to PCOS.

N.B: The diagnosis of PCO syndrome was made according to the Androgen Excess and Polycystic Ovarian Syndrome Society: the presence of the following criteria have been required for the diagnosis of PCO syndrome:

Hyperandrogenism: Hirsutism and/or Hyperandrogenaemia Ovarian Dysfunction : Oligo-Anovulation and /or Polycystic ovaries Exclusion of other Androgen Excess or related disorders as :( deficient nonclassic adrenal hyperplasia, androgen-secreting neoplasms, androgenic/anabolic drug use or abuse, Cushing's syndrome, the Hyperandrogenic-Insulin Resistance-Acanthosis Nigricans syndrome, thyroid dysfunction, and hyperprolactinemia).

Exclusion Criteria:

* Age below 20 or above 40. Women who intended to start a diet or a specific program of physical activity. Concurrent medical illness as cardiovascular, neoplastic and hepatic disorder. Pelvic pathology. Tubal, Uterine, Male factor of infertility. Endocrinological factors including: diabetes Mellitus,hypothyroidism, hyperprolactinaemia, Cushing's syndrome, and non- classical congenital adrenal hyperplasia.

Patients who are ovulatory during the ovarian cycle

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 85 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
pregnancy | 4 months
  polycystic ovarian syndrome patients getting pregnant on receiving Metformin

SECONDARY OUTCOMES:
Endometrial thickness and Sub Endometrial vascularity | 4 months
  Endometrial thickness and Sub Endometrial vascularity before and after receiving Metformin as markers of endometrial receptivity

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Khalaf, M.D, Principal Investigator — Ain Shams University Maternity Hospital
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided